CLINICAL TRIAL: NCT04570124
Title: Implementing the Systemic Treatment and Management of Postpartum Hypertension (STAMPP-HTN) Bundle in a High-risk Mississippi Population
Brief Title: STAMPP-HTN in a High-risk Rural Population of Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: University of Chicago (Other)
Responsible Party: Principal Investigator, Kedra Wallace, Associate Professor, PhD, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-0175
Record Dates: First submitted 2020-09-17; First posted 2020-09-30 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Hypertension in Pregnancy
Keywords: Hypertension; Blood Pressure; Post-Partum; Telemonitoring
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote Surveillance (Experimental): Women will use the home blood pressure monitoring device to record their blood pressure everyday for the first postpartum week, and then weekly until postpartum week 6.
  Interventions: Device: Home Blood Pressure Telemonitoring

INTERVENTIONS:
Device: Home Blood Pressure Telemonitoring — Women will complete a 9-question survey (pre-education) prior to discharge and will go over an education video a study team member. Once discharged, women will be asked to measure their blood pressure daily for the first postpartum week, and then weekly until postpartum week 6. Women who have a doctor's visit scheduled during the first 10 days, a member of the study team will meet them there to assess blood pressure and answer any questions. Women who do not have a visit scheduled they will have a telehealth visit during days 8-10 to complete the same assessments. At the final visit, participants will measure their blood pressure via HBPT, prior to returning the unit, complete a post-education questionnaire, a post-study questionnaire and have any questions or concerns addressed.

SUMMARY:
The purpose of this study is to determine if monitored blood pressure paired with education reduces maternal mortality and morbidity during the post-partum period in a high-risk rural population of women.

DETAILED DESCRIPTION:
Women with hypertension during pregnancy are at an increased risk of maternal mortality (death during or within 42 days of termination of pregnancy) and hypertension related morbidity. Black women, women with lower education and less access to health care resources also have increased maternal mortality and morbidity. This project will use Bluetooth enabled blood pressure devices to monitor blood pressure in a population of postpartum women at increased risk for maternal mortality and morbidity. We will compare the number of postpartum hypertensive incidences and severities to a population of women who did not have a postpartum blood pressure control intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent in a postpartum woman between 18-45 years of age at the time of study enrollment
2. Hospitalized for delivery with a hypertensive disorder of pregnancy as defined by ACOG 2019 Guidelines (chronic hypertension, HELLP syndrome, eclampsia, preeclampsia, gestational hypertension or new onset postpartum hypertension).
3. Ability to understand English or Spanish
4. Reliable access to the Internet and a Bluetooth mobile device
5. Willingness to download Omron Connect App and ability to use blood pressure monitor

Exclusion Criteria:

1. Does not meet Inclusion criteria
2. Postpartum or operative complication that prolongs hospital stay beyond postpartum day 10.
3. Patients who are currently participating in another clinical trial to evaluate a therapeutic intervention for control of blood pressure.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Determine if HBPT decreases the severity of postpartum hypertension complication | 9 months
  Postpartum outcomes between women being monitored to those from the previous year who received no postpartum blood pressure monitoring will be compared. Women will be monitored and we measure Systolic, Diastolic and Mean arterial pressure and to see if HPBT decreases the severity of postpartum hypertension from previous baseline measurements from women who had no interventions. Percentages of patients with controlled blood pressure at each time point will be compared to previous BP measurements.

SECONDARY OUTCOMES:
Increase awareness and knowledge of postpartum blood pressure control in a group of high-risk women | 9 months
  A 9-question survey will be given before any hypertension education is conducted with study participants and again at the end of the 6-week study. The pre-test and post-test will measure if women are more knowledgeable of how to monitor postpartum blood pressure. We will calculate test scores and knowledge based on increase or decrease of correct answers after participants received education and training.
Assess compliance using HBPT and adherence to blood pressure medication | 9 months
  Study completion records (per week) will be compared with study covariates (i.e. maternal race, age, parity). The measurement of compliance across different subcategories will determine what population, race and age group is most compliant. Percentage of women who are correctly taking medication will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Kedra Wallace, PhD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of MS Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Yes
All women will receive a de-identified laminated notecard that has their study results (Type of hypertensive pregnancy, gestational age at delivery, discharged and current blood pressure medication, last study blood pressure, and readmission status) on it that can be shared with any new provider (including non-obstetrical). As stated in the study consent, a letter outlining the same information will also be sent to the obstetrician listed in the patient's medical record
Supporting Information: CSR
Time Frame: Within 7 days of study completion each participant will receive their personal data as outlined in the study consent.
Access Criteria: Each patient will be mailed their information.

REFERENCES:
- [Derived] Moustafa ASZ, Yimer W, Perry A, Solis L, Belk S, Morris R, Spencer SK, Rana S, Wallace K. Report from a text-based blood pressure monitoring prospective cohort trial among postpartum women with hypertensive disorders of pregnancy. BMC Pregnancy Childbirth. 2024 May 3;24(1):340. doi: 10.1186/s12884-024-06511-1. PMID 38702619